CLINICAL TRIAL: NCT05489146
Title: Combining Transcranial Random Noise Stimulation and Functional Electrical Stimulation to Enhance Hand Function in Individuals With Chronic Stroke
Brief Title: t-RNS After Hand Recovery in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amit Sethi (Other)
Collaborators: Zynex Medical, Inc. (Industry); Neuroelectrics Corporation (Industry)
Responsible Party: Sponsor-Investigator, Amit Sethi, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO13090080
Record Dates: First submitted 2022-07-22; First posted 2022-08-05 (Actual); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Stroke
Keywords: stroke; hand; brain stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant, outcome assessor, investigator, and therapist providing the intervention were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- tRNS and FES facilitated task practice (Active Comparator): In this arm, participants received real transcranial random noise stimulation with FES facilitated task practice
  Interventions: Device: transcranial random noise stimulation and functional electrical stimulation facilitated task practice
- sham tRNS and FES facilitated task practice (Sham Comparator): In this arm, participants received sham transcranial random noise stimulation with FES facilitated task practice
  Interventions: Device: transcranial random noise stimulation and functional electrical stimulation facilitated task practice

INTERVENTIONS:
Device: transcranial random noise stimulation and functional electrical stimulation facilitated task practice — Participants were randomized to one of the two intervention groups [transcranial current stimulation (tRNS) and functional electrical stimulation (FES) or FES with sham tRNS] before pre-intervention testing. After randomization, participants underwent pre-intervention testing, followed by intervention 3 times per week for 6 weeks. Each intervention session lasted for 1 hour, where tRNS or sham-tRNS were delivered concurrently with the FES-facilitated task practice. tRNS or sham-tRNS was delivered for the first 30 minutes. Both tRNS and sham tRNS were delivered by the Starstim system. FES was delivered using the Neuromove system. All participants were treated by a licensed occupational therapist, who was trained on a manualized protocol.

SUMMARY:
Upper extremity (UE) paresis or weakness is one of the most frequent impairments after stroke. Despite intense rehabilitation, motor and functional recovery of patients with severe hand impairments is poor. Hence, there is a need for more effective treatments to enhance motor function in patients with severe hand impairments after stroke. Adaptive functional electrical stimulation (FES) appears to be a promising treatment and has the potential to facilitate active movement in individuals with severe impairments post-stroke. In addition, transcranial random noise stimulation (trns) is a widely studied, non-invasive and safe method to enhance the corticomotor excitability in individuals with chronic stroke. However, the effect of combining trns and adaptive FES in patients with severe hand impairments has not been investigated. Therefore, the purpose of this study is to investigate whether combining trns with FES will enhance hand function in individuals with chronic stroke than FES alone. The investigators predict that combining trns with FES will significantly enhance hand function than FES alone.

DETAILED DESCRIPTION:
The primary purpose of this study was to investigate whether combining transcranial random noise stimulation with functional electrical stimulation-facilitated task practice will enhance hand function in individuals with severe paresis post-stroke than functional electrical stimulation alone.

The study is an experimental randomized study comparing the effects of transcranial random noise stimulation with functional electrical stimulation to functional electrical stimulation alone on recovery of function in the more-affected hand in individuals with chronic stroke.

Participants were randomized to receive transcranial random noise stimulation and functional electrical stimulation-facilitated task practice or sham-transcranial random noise stimulation and functional electrical stimulation-facilitated task practice.

Participants received 18 treatment sessions over 6 weeks (3 times/week for 6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Episode (1 or more than one) of stroke at least 6 months prior
* Able to follow 3-step commands to rule out severe aphasia
* Unilateral hemiparesis
* Able to speak english
* No active drug or alcohol abuse, schizophrenia, other neurological or medical conditions that would confound results, or refractory depression
* Able to actively flex and extend the more-affected shoulder and elbow at least 30°.
* Able to elicit motor evoked potential in the flexor carpii radialis and extensor carpii radialis muscles of the affected hand.

Exclusion Criteria:

* Spasticity greater than equal to 2 on the Modified Ashworth Scale in shoulder, elbow, wrist and finger joints of the more-affected upper extremity
* Scores > 3 on the Amount scale of Motor Activity Log indicating good use of the more-affected hand
* Has ataxia determined via finger-to-nose testing section of the Fugl Meyer Upper Extremity assessment
* Has proprioceptive sensory deficits determined via a score of 2 on the position sense section (section H) of the Fugl Meyer Upper Extremity assessment proprioception
* Excessive pain > equal to 4 on Visual Analog Scale in the more-affected upper extremity
* Skin lesions on the more-affected upper extremity and scalp
* Individuals with implanted devices that may be affected by electrical stimulation
* Participating in concurrent therapy
* Individuals with seizures
* History of seizures, schizophrenia, Bipolar disorder (type I or II) [Answer yes to questions 16 and items of the (hypo) maniac module of MINI], current moderate, severe depression (Scores of >10 on PHQ-9) and other neurological or medical conditions that could confound results.
* Individuals with refractory depression, which are defined as individuals with severe depressive disorder that are resistant to antidepressants (Scores of >10 on PHQ-9).
* Current treatment with antipsychotics or benzodiazepines.
* Current treatment with bupropion, which may induce seizure.
* Scores < 24 on Mini Mental Status Examination
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sethi, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Neuromotor Recovery and Rehabilitation Lab, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.62 (10.69) | 54 (13.64) | 62.85 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Fugl Meyer Upper Extremity Scale [Mean (Standard Deviation); unit: score on a scale] — Fugl Meyer Upper Extremity Assessment (FMUE) measures motor impairment by asking the participant to perform various arm and hand motions. Items are scored on a 3-point ordinal scale, with 0 representing the inability to complete the item and 2 representing the ability to complete the item as asked. The minimum possible score of FMUE is 0, and the maximum score is 66, with a higher score indicating better performance.
  score on a scale | 28.5 (9.46) | 30.33 (12.27) | 29.28 (10.34)
Baseline Wolf Motor Function Test [Mean (Standard Deviation); unit: Seconds] — Wolf motor function test (WMFT) measures upper extremity motor ability through timed and functional tasks that increase in difficulty from simple UE movements requiring few degrees of freedom to tasks requiring the coordination of many degrees of freedom of movement. The WMFT is a 15-item test in which participants are given 2 minutes to complete each item. It measured in time with faster performance indicative of better UE motor control.
  Seconds | 41.88 (33.07) | 49.32 (29.43) | 45.07 (30.60)
Baseline Grip Strength [Mean (Standard Deviation); unit: Pounds] — Grip strength is measured with a hand-held dynamometer. The participant will do three trials and then take the average score. The average score is compared to age and gender-matched standardized scores.
  Pounds | 12.90 (7.46) | 13.15 (6.89) | 13.01 (6.94)
Baseline of Hand Subscale of Stroke Impact Scale [Mean (Standard Deviation); unit: score on a scale] — The Stroke Impact Scale measures the impact of stroke on the participant's health and daily life. It is a self-report measure, and each item is scored on a 5-item Likert scale. We completed items from the hand subscale. The minimum possible score is 5, and the maximum score is 25 with a higher score indicative of better recovery.
  score on a scale | 9.75 (3.92) | 11.17 (2.64) | 10.35 (3.38)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fugl Meyer Upper Extremity Scale at Post Treatment
Description: Fugl Meyer Upper Extremity Scale (FMUE) is considered the gold standard in upper extremity rehabilitation trials and measures upper extremity motor control by asking the participant to perform various arm and hand motions. Items are scored on a 3-point ordinal scale with 0 representing inability to complete the item and 2 representing the ability to complete the item as asked. We will use the total score, which ranges from 0-66. Higher score suggest better upper extremity motor control. The FMUE has been shown to have good reliability and validity.
Time Frame: Baseline, 6 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 8 | 6
score on a scale | 35.25 (4.27) | 33.5 (3.83)
Statistical Analysis 1: Comparison: tRNS and FES Facilitated Task Practice vs Sham tRNS and FES Facilitated Task Practice; Test type: Superiority; p = 0.046, Mixed Models Analysis

2. Primary Outcome: Change From Baseline in Fugl Meyer Upper Extremity Scale at 3 Months Post Treatment
Description: as for outcome 1
Time Frame: Baseline, 3 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 8 | 6
score on a scale | 37.25 (4.73) | 33.5 (4.68)
Statistical Analysis 1: Comparison: tRNS and FES Facilitated Task Practice vs Sham tRNS and FES Facilitated Task Practice; Test type: Superiority; p = 0.003, Mixed Models Analysis

3. Secondary Outcome: Change From Baseline in Wolf Motor Function Test at Post Treatment
Description: The Wolf Motor Function Test (WMFT) is a 15-item test in which participants are given 2 minutes to complete each item. The items increase in difficulty from simple UE movements requiring few degrees of freedom (e.g. placing hand on a table) to tasks requiring the coordination of many degrees of freedom of movement (e.g. folding a towel). We used average time taken to complete the 15-items. Faster performance is indicative of better task performance. The WMFT is a valid and reliable test of UE function post-stroke.
Time Frame: Baseline, 6 weeks.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 8 | 6
Seconds | 33.46 (9.24) | 42.79 (13.58)
Statistical Analysis 1: Comparison: tRNS and FES Facilitated Task Practice vs Sham tRNS and FES Facilitated Task Practice; Test type: Superiority; p > 0.05, Mixed Models Analysis

4. Secondary Outcome: Change From Baseline in Wolf Motor Function Test at 3 Months Post Treatment
Description: as for outcome 3
Time Frame: Baseline, 3 months.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 8 | 6
Seconds | 34.18 (10.52) | 37.38 (12.13)
Statistical Analysis 1: Comparison: tRNS and FES Facilitated Task Practice vs Sham tRNS and FES Facilitated Task Practice; Test type: Superiority; p > 0.05, ANCOVA

5. Secondary Outcome: Change From Baseline in Grip Strength at Post Treatment
Description: Grip strength measures the amount of maximum voluntary grip force of the weak hand using a hand-held dynamometer. We will use the maximum amount of force in pounds.
Time Frame: Baseline, 6 weeks.
Measure: Mean (Standard Error); unit: Pounds
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 8 | 6
Pounds | 17.50 (5.53) | 15.60 (3.21)
Statistical Analysis 1: Comparison: tRNS and FES Facilitated Task Practice vs Sham tRNS and FES Facilitated Task Practice; Test type: Superiority; p > 0.05, Mixed Models Analysis

6. Secondary Outcome: Change From Baseline in Grip Strength at 3 Months Post Treatment
Description: as for outcome 5
Time Frame: Baseline, 3 months.
Measure: Mean (Standard Error); unit: Pounds
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 8 | 6
Pounds | 16.49 (3.98) | 16.19 (4.11)
Statistical Analysis 1: Comparison: tRNS and FES Facilitated Task Practice vs Sham tRNS and FES Facilitated Task Practice; Test type: Superiority; p > 0.05, Mixed Models Analysis

7. Secondary Outcome: Change From Baseline in Hand Subscale of Stroke Impact Scale at Post Treatment
Description: The Hand sub scale of Stroke Impact Scale 3.0 (HSIS) will be used to measure the impact of stroke on participants' health and daily life. The Hand sub scale SIS is a self-report measure, which evaluates the ability of the hand to participate in daily tasks. The scale consists of 5 items and each item is scored on a 5-item Likert scale. We will use the total score, which ranges from 1-25, with a higher score indicative of better recovery.
Time Frame: Baseline, 6 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 8 | 6
score on a scale | 15.88 (1.47) | 12.17 (1.92)
Statistical Analysis 1: Comparison: tRNS and FES Facilitated Task Practice vs Sham tRNS and FES Facilitated Task Practice; Test type: Superiority; p = 0.001, Mixed Models Analysis

8. Secondary Outcome: Change From Baseline in Hand Subscale of Stroke Impact Scale at 3 Months Post Treatment
Description: as for outcome 7
Time Frame: Baseline, 3 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 8 | 6
score on a scale | 14.38 (1.63) | 12.67 (1.94)
Statistical Analysis 1: Comparison: tRNS and FES Facilitated Task Practice vs Sham tRNS and FES Facilitated Task Practice; Test type: Superiority; p = 0.035, Mixed Models Analysis

9. Secondary Outcome: Change From Baseline in Action Research Arm Test at Post Treatment
Description: Action Research Arm Test (ARAT) measures arm and hand recovery after stroke. The ARAT is a 19-item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). The total score from the 4 sub-tests ranges from 0-57. We will use total score. Higher scores suggest better ability to grasp, grip and perform arm movements.
Time Frame: Baseline, 6 weeks.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Action Research Arm Test at 3 Months Post Treatment
Description: as for outcome 9
Time Frame: Baseline, 3 months.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Baseline in H-reflex at Post Treatment
Description: H-reflex testing will be used to record the spastic reflex in the Flexor carper radials (FCR) muscle of the weak hand. H-reflex is the reflex reaction of the muscles after electrical stimulation of the peripheral nerves supplying the muscle. Here we will stimulate the median nerve to stimulate and record the H-reflex values of the H-reflex. Normalized H-reflex values will be used. Lower values represent decrease in spasticity in the FCR after treatment.
Time Frame: Baseline, 6 weeks.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Baseline in H-reflex at 3 Months Post Treatment
Description: as for outcome 11
Time Frame: Baseline, 3 weeks.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Baseline in Brain Activity at Post Treatment
Description: Electroencephalography (EEG) will be used to record brain activity. EEG will be recorded while the participant is attempting to perform movements of the weak hand, or while they are at rest. We will attach EEG sensors to the scalp to measure brain activity. We will compute power of the EEG signal in the alpha and beta bands. Higher values will represent increase in brain activity post treatment.
Time Frame: Baseline, 6 weeks.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Baseline in Brain Activity at 3 Months Post Treatment
Description: as for outcome 13
Time Frame: Baseline, 3 months.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change in Baseline in Muscle Activity at Post Treatment
Description: We will record muscle activity using Electromyography (EMG). We will collect EMG using 2 methods: basic EMG and High Definition EMG. In the basic EMG we will use (2 sensors) for the extensor carpi radials and flexor carp radials muscles and record muscle activity during wrist movements. In the High Definition EMG participants will wear a forearm sleeve, which will allows us to collect activity from multiple muscles, responsible for grasping and releasing objects of daily use. We will calculate the max voluntary contraction of the forearm muscles. Normalized values will be used. Higher values will represent increased muscle activity post treatment.
Time Frame: Baseline, 6 weeks.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change in Baseline in Muscle Activity at 3 Months Post Treatment
Description: as for outcome 15
Time Frame: Baseline, 3 months.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change in Baseline in Brain Excitability at Post Treatment
Description: We will use Transcranial Magnetic Stimulation (TMS) to measures the excitability of motor pathways in the brain. Normalized values will used. Higher values represent higher brain excitability post treatment.
Time Frame: Baseline, 6 weeks.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change in Baseline in Brain Excitability at 3 Months Post Treatment
Description: as for outcome 17
Time Frame: Baseline, 3 months.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Change in in Baseline in Upper Extremity Kinematics at Post Treatment
Description: We will use motion capture system to measure changes in upper extremity kinematics, including shoulder, elbow, wrist joint range of motion. The values will be measured in degrees. Higher values will represent greater range of motion post treatment.
Time Frame: Baseline, 6 weeks.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change in in Baseline in Upper Extremity Kinematics at 3 Months Post Treatment
Description: as for outcome 19
Time Frame: Baseline, 3 months.
Population: Data was not collected because of the feasibility of testing or participants' burden.
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event was collected before and after each 1-hour treatment session, 3 times per week for 6 weeks
Arm/Group | tRNS and FES Facilitated Task Practice | Sham tRNS and FES Facilitated Task Practice
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT05489146/Prot_SAP_000.pdf